CLINICAL TRIAL: NCT00439686
Title: A Phase IB/IIA Study of the Saftey and Activity of Intravenous Isophosporamide Mustard (ZIO-201) in Patients With Advanced Sarcoma
Brief Title: Study of ZIO-201 in Advanced Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Alaunos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPM2001
Record Dates: First submitted 2007-02-22; First posted 2007-02-26 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Sarcoma
MeSH Terms: interventions — palifosfamide lysine

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: ZIO-201

INTERVENTIONS:
Drug: ZIO-201 — ZIO-201 given for 3 consecutive days to be repeated every 21 days for up to 6 months

SUMMARY:
The study of safety of Isophosphoramide Mustard (IPM) in the treatment of advanced sarcoma.

ELIGIBILITY:
Metastatic and /or unresectable disease state after previous standard chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2006-02; Primary Completion 2008-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
toxicities | 6 months

SECONDARY OUTCOMES:
pharmacokinetics | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Lewis, MD, PhD, Study Director — ZIOPHARM Oncology, Inc
Locations (2):
- United States (2):
  - Santa Monica, California
  - Ann Arbor, Michigan